CLINICAL TRIAL: NCT05497999
Title: Racial Inequality in Inhaler Fills for COPD - A Trial of Reduced Cost-Sharing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Humana Co.Ltd. (Industry)
Responsible Party: Principal Investigator, Sumit Agarwal, Instructor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0916
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Cost sharing; Health insurance; Inhalers; Adherence; Disparities
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): With Black and White Subgroups
  Interventions: Other: Proactive Outreach
- Control Group (Active Comparator): With Black and White Subgroups
  Interventions: Other: No Proactive Outreach

INTERVENTIONS:
Other: Proactive Outreach — The treatment is proactive outreach that sought to enroll individuals in a VBID program available to all enrollees that provided: 1) large reductions in cost-sharing for maintenance inhalers, and 2) telephone-based COPD medication management services.
  Proactive outreach for those randomized to the treatment arm included, at a minimum, a phone call and letter in the mail from Humana. Proactive outreach could also have included an email, text message, and/or provider referral.
  Arms: Treatment Group
Other: No Proactive Outreach — Control group participants received no proactive outreach but could call to enroll themselves in the VBID program if they learned about it through traditional means, such as the benefits description manual.
  Arms: Control Group

SUMMARY:
In partnership with a large Medicare Advantage (MA) insurer (Humana, Inc.) and as part of a Center for Medicare and Medicaid Innovation demonstration program of Value-Based Insurance Design (VBID), the investigators propose to study a randomized controlled quality improvement trial in which Humana randomized MA beneficiaries with COPD to receive proactive outreach for a VBID benefit that provided large reductions in cost-sharing for their maintenance inhalers and telephone-based COPD medication management services in 2020 and 2021. The investigators will analyze changes in racial disparities for inhaler fills, clinical outcomes, health care spending, and acute care utilization.

ELIGIBILITY:
Inclusion Criteria:

* Has COPD diagnosis
* Receives health services and prescription drug benefits through a Humana Medicare Advantage plan that includes Part D coverage
* Has at least one prior fill of a COPD maintenance inhaler in the prior 12 months
* Not fully adherent to maintenance inhaler (PDC < 80%) in year prior to randomization

Exclusion Criteria:

* Enrolled in Part D Low-Income Subsidy program
* On hospice
* Has end-stage renal disease
* Has mild COPD (i.e., COPD diagnosis but no maintenance inhaler fill, no pulmonary function tests in year prior year, and no acute care use for COPD)
* Enrolled in Humana plan for less than 3 months
* In the coverage gap phase of MA plan at time of assignment
* Receives primary care at select locations of Humana subsidiaries (CenterWell or Conviva)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19113 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Maintenance inhaler adherence | 1 Year
  A maintenance inhaler is defined as any inhaler with an inhaled corticosteroid, long-acting beta-agonist, and/or long-acting antimuscarinic antagonist. The proportion of days covered (PDC), a common claims-based measure of adherence, is calculated by dividing number of days covered by a prescription by the total number of days eligible for the medication. In constructing the measure, days covered (numerator) will be number of days on any maintenance inhaler (whether one of a single class, multiple of differing classes, or changes between inhalers), and the days eligible (denominator) will be number of days in the observation period. The primary analysis will treat PDC as a continuous measure.

SECONDARY OUTCOMES:
Frequency of acute moderate-to-severe exacerbations | 1 Year
  An exacerbation is defined as any acute worsening of symptoms that requires antibiotics or systemic steroids. Moderate exacerbations are those that do not result in hospitalization or death and therefore captures those exacerbations treated on an outpatient basis. Severe exacerbations are exacerbations that result in hospitalization.
Number of short-acting inhaler filled | 1 Year
  A short-acting inhaler is defined as any inhaler with a short-acting beta agonist and/or short-acting antimuscarinic antagonist.
Total spending | 1 Year
  Total spending includes both the insurer's payments and beneficiary's out-of-pocket payments over the course of the calendar year. It includes spending across types of service (e.g., drugs) and settings (e.g., acute care).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - Humana, Inc., Louisville, Kentucky
  - Harvard Medical School, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agarwal SD, Metzler E, Chernew M, Thomas E, Press VG, Boudreau E, Powers BW, McWilliams JM. Reduced Cost Sharing and Medication Management Services for COPD: A Randomized Clinical Trial. JAMA Intern Med. 2024 Oct 1;184(10):1186-1194. doi: 10.1001/jamainternmed.2024.3499. PMID 39073823

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT05497999/Prot_SAP_000.pdf